CLINICAL TRIAL: NCT05649540
Title: Optimization of Vonoprazan-based Dual Therapy for Helicobacter Pylori:a Prospective, Multicenter, Open Label, Randomized Controlled Study:
Brief Title: Optimization of Vonoprazan-based Dual Therapy for Helicobacter Pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Director of Gastroenterology, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20221124-07
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; dual therapy; eradication rate; safety; microbiota
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high dose amoxicillin with vonoprazan group (Active Comparator): vonoprazan 20mg bid and amoxicillin 1000mg tid for 14 days
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin
- standard dose amoxicillin with vonoprazan group (Experimental): vonoprazan 20mg bid and amoxicillin 1000mg bid for 14 days
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin
- low dose amoxicillin with vonoprazan group (Experimental): vonoprazan 20mg bid and amoxicillin 500mg tid for 14 days
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin

INTERVENTIONS:
Drug: Vonoprazan — Potassium-competitive acid blocker
Drug: Amoxicillin — Antibiotic for H. pylori eradication

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of vonoprazan with different doses of amoxicillin for Helicobacter Pylori.

DETAILED DESCRIPTION:
This study intends to select the patients with Hp infection in 13 tertiary hospitals across our country, and randomly give the three therapies to compare the eradication rate, compliance, the rate of adverse events, so as to provide some advices for the selection of appropriate eradication therapy, then collect an efficient, convenient and safe therapy for patients with H.pylori infection.

Before receiving the treatment plan, general information and relevant medical history of the subjects were collected through electronic questionnaires.The experimental data will be collected and recorded through follow-up by phone or WeChat during the experiment.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18 and 70 years; Sexes eligible for study: both;
2. patients who are diagnosed with Helicobacter pylori with 13C urea breath test or 14C urea breath test;
3. treatment-naive patients or patients who failed to eradicate Helicobacter pylori in the past but haven't undergone eradication therapy in the past six months;
4. voluntary to be involved in the study and written informed consent was obtained from all patients

Exclusion Criteria:

1. allergic reactions to the study drugs;
2. patients with peptic ulcer;
3. patients who underwent eradication therapy for Helicobacter pylori during the last six months;
4. patients who took antibiotics,bismuth agents,probiotics within four weeks prior to treatment and those who took H2 receptor antagonists,proton pump inhibitors(PPIs) or potassium competitive acid blockers within two weeks prior to treatment;
5. patients who are taking glucocorticoids, non-steroidal anti-inflammatory drugs or anticoagulants;
6. patients who have history of esophageal or gastric surgery;
7. pregnant or lactating women;
8. patients who have severe concurrent diseases such as hepatic,cardiovascular,respiratory,renal disorders or malignancies;
9. Alcohol abusers
10. MALT lymphoma of stomach or malignant tumor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-07-06 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | four to eight weeks after completion of the medication
  Helicobacter pylori Eradication will be determined by ¹³C-urea breath test four to six weeks after completion of the medication. The eradication rates will be evaluated by intention-to-treat (ITT) and per-protocol (PP) analysis.

SECONDARY OUTCOMES:
Adverse event | Within 7 days after completion of therapy
  Adverse drug reactions are classified into six types: dose-related, non-dose-related, dose-related and time-related, time-related, withdrawal, and failure of therapy.
Compliance Rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication
Microbiota influence | baseline, within 1 day after completion of therapy, Within 6 weeks after completion of therapy
  Collect the tongue coating and feces of some patients for flora analysis

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Zhang, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (13):
- China (13):
  - Changshu No.1 People's Hospital, Changshu, Jiangsu
  - Changzhou Traditional Chinese Medicine Hospital, Changzhou, Jiangsu
  - The first people's hospital of Lianyungang, Lianyungang, Jiangsu
  - Jiangsu Province Hospital on Integration of Chinese and Western Medicine, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Jiangbei Hospital, Nanjing, Jiangsu
  - Sir Run Run Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Taixing People's Hospital, Taishing, Jiangsu
  - The Fourth People's Hospital of Taizhou, Taizhou, Jiangsu
  - The First People's Hospital of Xuzhou, Xuzhou Municipal Hospital Affiliated to Xuzhou Medical University, Xuzhou, Jiangsu
  - Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu
  - The Affiliated Zhangjiagang Hospital of Soochow University, Zhangjiagang, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sugano K, Tack J, Kuipers EJ, Graham DY, El-Omar EM, Miura S, Haruma K, Asaka M, Uemura N, Malfertheiner P; faculty members of Kyoto Global Consensus Conference. Kyoto global consensus report on Helicobacter pylori gastritis. Gut. 2015 Sep;64(9):1353-67. doi: 10.1136/gutjnl-2015-309252. Epub 2015 Jul 17. PMID 26187502
- [Background] Malfertheiner P, Megraud F, Rokkas T, Gisbert JP, Liou JM, Schulz C, Gasbarrini A, Hunt RH, Leja M, O'Morain C, Rugge M, Suerbaum S, Tilg H, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study group. Management of Helicobacter pylori infection: the Maastricht VI/Florence consensus report. Gut. 2022 Aug 8:gutjnl-2022-327745. doi: 10.1136/gutjnl-2022-327745. Online ahead of print. PMID 35944925
- [Background] Ford AC, Malfertheiner P, Giguere M, Santana J, Khan M, Moayyedi P. Adverse events with bismuth salts for Helicobacter pylori eradication: systematic review and meta-analysis. World J Gastroenterol. 2008 Dec 28;14(48):7361-70. doi: 10.3748/wjg.14.7361. PMID 19109870
- [Background] Gao CP, Zhang D, Zhang T, Wang JX, Han SX, Graham DY, Lu H. PPI-amoxicillin dual therapy for Helicobacter pylori infection: An update based on a systematic review and meta-analysis. Helicobacter. 2020 Aug;25(4):e12692. doi: 10.1111/hel.12692. Epub 2020 Apr 20. PMID 32314468
- [Background] Furuta T, Shirai N, Kodaira M, Sugimoto M, Nogaki A, Kuriyama S, Iwaizumi M, Yamade M, Terakawa I, Ohashi K, Ishizaki T, Hishida A. Pharmacogenomics-based tailored versus standard therapeutic regimen for eradication of H. pylori. Clin Pharmacol Ther. 2007 Apr;81(4):521-8. doi: 10.1038/sj.clpt.6100043. Epub 2007 Jan 10. PMID 17215846
- [Background] Guan JL, Hu YL, An P, He Q, Long H, Zhou L, Chen ZF, Xiong JG, Wu SS, Ding XW, Luo HS, Li PY. Comparison of high-dose dual therapy with bismuth-containing quadruple therapy in Helicobacter pylori-infected treatment-naive patients: An open-label, multicenter, randomized controlled trial. Pharmacotherapy. 2022 Mar;42(3):224-232. doi: 10.1002/phar.2662. Epub 2022 Feb 5. PMID 35075679
- [Derived] Peng R, Cai P, Zhang Z, Lv S, Chen G, Xu Y, He B, Sun M, Dai X, Yan K, Shen L, Wang J, Li W, Yin R, Ge J, Hu D, Hu K, Xu X, Li H, Pan C, Duan Z, Gao X, Zhang Z, Liu W. Efficacy of Three Amoxicillin Doses in Vonoprazan Dual Therapy for Helicobacter pylori Eradication: A Randomized Noninferiority Trial. Helicobacter. 2025 May-Jun;30(3):e70050. doi: 10.1111/hel.70050. PMID 40481714